CLINICAL TRIAL: NCT01559220
Title: Deep Brain Stimulation (DBS) for Treatment of the Cognitive, Behavioral, and Functional Disability of Alzheimer's Disease
Brief Title: Deep Brain Stimulation for the Treatment of Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Rezai, MD (Other)
Responsible Party: Sponsor-Investigator, Ali Rezai, MD, MD, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2011H0362
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Open Label (Experimental): DBS Implant and stimulation
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Implanted device
  Other Names: Deep Brain Stimulation Device

SUMMARY:
The purpose of this clinical study is to investigate the safety and efficacy of deep brain stimulation (DBS)as a treatment option for patients with cognitive, behavioral, and functional disability of Alzheimer's disease.

DETAILED DESCRIPTION:
Open label pilot study

* Expected direct benefit on the modulation of neuronal networks.
* Expected indirect benefit via potential enhancements of memory, executive functions, cognition behavioral control, and functional abilities.

Up to 10 subjects will be implanted with bilateral DBS systems, participants are expected to be on study for about 23 months.

* Develop a multidisciplinary clinical research protocol to evaluate the efficacy of ventral striatum, nucleus accumbens, and internal capsule for the amelioration of disability caused by Alzheimer's Disease.
* Enroll up to 10 patients into an open label study to evaluate the safety and efficacy of DBS for Alzheimer's Disease patients with mild to moderate disability.
* Determine an initial DBS titration and stimulation settings protocol for use in subsequent controlled trials.
* Evaluate the outcomes of this study based on clinical, laboratory, biomarker, imaging, cognitive, behavioral, and functional assessments.
* Determine what domains of cognitive, behavioral and functioning impairment show the greatest response to DBS.
* Examine the potential benefit of stimulation combined with behavioral and rehabilitation interventions in comparison to stimulation alone.
* Evaluate the influence of DBS on physiological and functional changes in cortical and subcortical networks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD according to the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria

Exclusion Criteria:

* Has significant neurological disease, other than Alzheimer's disease, e.g., multiple sclerosis, Parkinson's disease and ischemic stroke, or severe brain atrophy or the presence of subdural hygromas or subdural hematomas.
* Evidence of substance abuse (alcohol or other drug) abuse or dependence during the previous 12 months (DSM-IV Criteria).

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Clinical Dementia Rating Scale | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezai, MD, Principal Investigator — Ohio State University
Locations (1):
- Wexner Medical Center at the Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No